CLINICAL TRIAL: NCT05468788
Title: Evaluating the Use of Theatre to Decrease Depression and Anxiety Among Adolescents With Chronic Medical Conditions (CMCs)
Brief Title: Theatre in Adolescents With Chronic Medical Conditions (CMCs)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants were recruited to conduct a randomized controlled trial.
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-0322
Record Dates: First submitted 2022-07-12; First posted 2022-07-21 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: One group will receive a new behavioral intervention; the other group will receive improvisational theatre alone
Who Masked: Participant
Masking Description: The participants will not know which group they are in, as they will not be familiar with the particular procedure of the intervention being studied
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrative Community Therapy (ICT) Intervention Arm (Experimental): Participants will perform scenes related to having a chronic medical condition and they will be guided through conversations about their feelings and coping methods.
  Interventions: Behavioral: Intervention: Integrative Community Therapy-based Psychodrama
- Improvisational Theatre Arm (Sham Comparator): Participants will perform generic improvisational theatre with no instruction on feelings or coping methods.
  Interventions: Behavioral: Control: Improvisational Theatre

INTERVENTIONS:
Behavioral: Intervention: Integrative Community Therapy-based Psychodrama — Participants produce theatre scenes depicting issues that they have experienced. Group leaders then use a guide to facilitate a discussion of participants' feelings, coping strategies, and sharing of local knowledge.
  Other Names: Intervention: ICT-based Psychodrama
  Arms: Integrative Community Therapy (ICT) Intervention Arm
Behavioral: Control: Improvisational Theatre — Participants play improvisational theatre games.
  Arms: Improvisational Theatre Arm

SUMMARY:
Investigators are building a program that uses improvisation to teach kids and teens with medical issues healthy ways to cope. Medical issues have been linked to anxiety and depression. Doing theatre can prevent these complications. Participants will meet in groups of about ten for ten weeks to do improvisation that is fun and supportive. Participants will meet with a study team member before the program starts, after the program ends, six months after the program ends, and twelve months after the program ends. At these visits, participants will be screened for anxiety, depression, quality of life, and will be given a short interview.

DETAILED DESCRIPTION:
Adolescents with chronic medical conditions are at increased risk for anxiety and depression compared to other people their age. Therapies that use role-play prevent anxiety and depression. However, often these studies do not have an underlying psychological framework, or there is not enough information to replicate the program. Investigators designed an intervention using role-play based on Integrative Community Therapy, developed in the 1980s by Dr. Adalberto Barreto. This program will help adolescents with chronic medical conditions explore their feelings about issues related to having a chronic condition, learn new coping strategies, and help one another find support among peers.

This treatment will take place once a week for 10 weeks and investigators will compare the effects to those derived from improvisational theatre alone. To evaluate this new treatment, the study team will screen participants for anxiety, depression, quality of life, and will give a short qualitative interview. This will occur before and after the intervention, 6 months after the intervention, and 1 year after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Identify as having a CMC
* In grades kindergarten to 12th grade during the year recruited for the study

  * 5 years of age and ≤ 19 years of age at the start of the intervention
* Able and willing to participate in improvisational theatre in spoken English
* Able to understand and answer standard questionnaires used for evaluation in English (with or without accommodation)

Exclusion Criteria:

* None

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety and Depression | Baseline to 10 weeks
  Anxiety and Depression as evaluated by the Revised Children's Anxiety and Depression Scale; Scored 0-30; higher score indicates worse outcome
Anxiety and Depression | Baseline to 6 months
  Anxiety and Depression as evaluated by the Revised Children's Anxiety and Depression Scale; Scored 0-30; higher score indicates worse outcome
Anxiety and Depression | Baseline to 12 months
  Anxiety and Depression as evaluated by the Revised Children's Anxiety and Depression Scale; Scored 0-30; higher score indicates worse outcome
Disease-Related Quality of Life | Baseline to 10 weeks
  Disease-Related Quality of Life as evaluated by Qualitative Interview
Disease-Related Quality of Life | Baseline to 6 months
  Disease-Related Quality of Life as evaluated by Qualitative Interview
Disease-Related Quality of Life | Baseline to 12 months
  Disease-Related Quality of Life as evaluated by Qualitative Interview
Disease-Related Quality of Life | Baseline to 10 weeks
  Disease-Related Quality of Life as evaluated by Pediatric Quality of Life Inventory; Scored 0-100; higher score indicates better outcome
Disease-Related Quality of Life | Baseline to 6 months
  Disease-Related Quality of Life as evaluated by Pediatric Quality of Life Inventory; Scored 0-100; higher score indicates better outcome
Disease-Related Quality of Life | Baseline to 12 months
  Disease-Related Quality of Life as evaluated by Pediatric Quality of Life Inventory; Scored 0-100; higher score indicates better outcome
Knowledge and Utilization of Coping Strategies | Baseline to 10 weeks
  Knowledge and Utilization of Coping Strategies as evaluated by Qualitative Interview
Knowledge and Utilization of Coping Strategies | Baseline to 6 months
  Knowledge and Utilization of Coping Strategies as evaluated by Qualitative Interview
Knowledge and Utilization of Coping Strategies | Baseline to 12 months
  Knowledge and Utilization of Coping Strategies as evaluated by Qualitative Interview
Knowledge and Utilization of Coping Strategies | Baseline to 10 weeks
  Knowledge and Utilization of Coping Strategies as evaluated by KidCope Checklist; Scored 0-120; higher score indicates better outcome
Knowledge and Utilization of Coping Strategies | Baseline to 6 months
  Knowledge and Utilization of Coping Strategies as evaluated by KidCope Checklist; Scored 0-120; higher score indicates better outcome
Knowledge and Utilization of Coping Strategies | Baseline to 12 months
  Knowledge and Utilization of Coping Strategies as evaluated by KidCope Checklist; Scored 0-120; higher score indicates better outcome
Empathy | Baseline to 10 weeks
  Empathy as evaluated by Qualitative Interview
Empathy | Baseline to 6 months
  Empathy as evaluated by Qualitative Interview
Empathy | Baseline to 12 months
  Empathy as evaluated by Qualitative Interview

CONTACTS AND LOCATIONS:
Overall Officials: Karen A Ephlin, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Primary Care South Wilkes-Barre, Wilkes-Barre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young KS, Sandman CF, Craske MG. Positive and Negative Emotion Regulation in Adolescence: Links to Anxiety and Depression. Brain Sci. 2019 Mar 29;9(4):76. doi: 10.3390/brainsci9040076. PMID 30934877
- [Background] Jones LC, Mrug S, Elliott MN, Toomey SL, Tortolero S, Schuster MA. Chronic Physical Health Conditions and Emotional Problems From Early Adolescence Through Midadolescence. Acad Pediatr. 2017 Aug;17(6):649-655. doi: 10.1016/j.acap.2017.02.002. Epub 2017 Feb 12. PMID 28215656
- [Background] Cobham VE, Hickling A, Kimball H, Thomas HJ, Scott JG, Middeldorp CM. Systematic Review: Anxiety in Children and Adolescents With Chronic Medical Conditions. J Am Acad Child Adolesc Psychiatry. 2020 May;59(5):595-618. doi: 10.1016/j.jaac.2019.10.010. Epub 2019 Oct 30. PMID 31676391
- [Background] Compas BE, Jaser SS, Dunn MJ, Rodriguez EM. Coping with chronic illness in childhood and adolescence. Annu Rev Clin Psychol. 2012;8:455-80. doi: 10.1146/annurev-clinpsy-032511-143108. Epub 2011 Dec 20. PMID 22224836
- [Background] Greenberg MT, Weissberg RP, O'Brien MU, Zins JE, Fredericks L, Resnik H, Elias MJ. Enhancing school-based prevention and youth development through coordinated social, emotional, and academic learning. Am Psychol. 2003 Jun-Jul;58(6-7):466-74. doi: 10.1037/0003-066x.58.6-7.466. PMID 12971193
- [Background] Hersov L. Psychotherapy for Children and Adolescents. Evidence-based Treatments and Case Examples. Child Adolesc Ment Health. 2006 May;11(2):124-125. doi: 10.1111/j.1475-3588.2006.00399_5.x. No abstract available. PMID 32811094
- [Background] Feniger-Schaal R, Koren-Karie N. Using Drama Therapy to Enhance Maternal Insightfulness and Reduce Children's Behavior Problems. Front Psychol. 2021 Jan 20;11:586630. doi: 10.3389/fpsyg.2020.586630. eCollection 2020. PMID 33551907
- [Background] Blacker J, Watson A, Beech AR. A combined drama-based and CBT approach to working with self-reported anger aggression. Crim Behav Ment Health. 2008;18(2):129-37. doi: 10.1002/cbm.686. PMID 18383198
- [Background] Joronen K, Hakamies A, Astedt-Kurki P. Children's experiences of a drama programme in social and emotional learning. Scand J Caring Sci. 2011 Dec;25(4):671-8. doi: 10.1111/j.1471-6712.2011.00877.x. Epub 2011 Mar 1. PMID 21362006
- [Background] Daykin N, Orme J, Evans D, Salmon D, McEachran M, Brain S. The impact of participation in performing arts on adolescent health and behaviour: a systematic review of the literature. J Health Psychol. 2008 Mar;13(2):251-64. doi: 10.1177/1359105307086699. PMID 18375630
- [Background] Joronen K, Rankin SH, Astedt-Kurki P. School-based drama interventions in health promotion for children and adolescents: systematic review. J Adv Nurs. 2008 Jul;63(2):116-31. doi: 10.1111/j.1365-2648.2008.04634.x. PMID 18537845
- [Background] Miranda NA, Berardinelli LM, Saboia VM, Brito ID, Santos RD. Interdisciplinary care praxis in groups of people living with fibromyalgia. Rev Bras Enferm. 2016 Nov-Dec;69(6):1115-1123. doi: 10.1590/0034-7167-2016-0279. English, Portuguese. PMID 27925088
- [Background] Weigensberg MJ, Vigen C, Sequeira P, Spruijt-Metz D, Juarez M, Florindez D, Provisor J, Peters A, Pyatak EA. Diabetes Empowerment Council: Integrative Pilot Intervention for Transitioning Young Adults With Type 1 Diabetes. Glob Adv Health Med. 2018 Mar 8;7:2164956118761808. doi: 10.1177/2164956118761808. eCollection 2018. PMID 29552422
- [Background] Chorpita BF, Yim L, Moffitt C, Umemoto LA, Francis SE. Assessment of symptoms of DSM-IV anxiety and depression in children: a revised child anxiety and depression scale. Behav Res Ther. 2000 Aug;38(8):835-55. doi: 10.1016/s0005-7967(99)00130-8. PMID 10937431
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Spirito A, Stark LJ, Williams C. Development of a brief coping checklist for use with pediatric populations. J Pediatr Psychol. 1988 Dec;13(4):555-74. doi: 10.1093/jpepsy/13.4.555. No abstract available. PMID 3216277